CLINICAL TRIAL: NCT03698279
Title: Safety and Immunogenicity of Different Dosages of High-Dose Quadrivalent Influenza Vaccine in Children 6 Months to 17 Years of Age
Acronym: QHD04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: QHD04; U1111-1189-3713 (Other: WHO); 2018-005026-39 (EudraCT Number)
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Results first posted 2020-06-01 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Antigens, Surface

STUDY DESIGN:
Intervention Model Description: The study was divided into 13 groups and enrolled participants in 4 stages. The study used a stepwise age de-escalation and dose ascension design for children 6 months to less than (<) 5 years of age.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Modified double-blind: the participant's parent / legally acceptable representative, the Investigator, and other study personnel remained unaware of the treatment assignments throughout the trial. An unblinded vaccine administrator administered the appropriate vaccine but was not involved in safety data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1: QIV-HD 30 μg (US: 6 months to 17 years) (Experimental): Participants from United States (US) (aged 6 months to 17 years) received single injection of 30 microgram (μg) QIV-HD, intramuscularly (IM) at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 30 μg (split-virion, inactivated)
- Group 2: QIV-HD 45 μg (US: 6 months to 17 years) (Experimental): Participants from US (aged 6 months to 17 years) received single injection of 45 μg QIV-HD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 45 μg, (split-virion, inactivated)
- Group 3: QIV-HD, 60 μg (US: 6 months to 17 years) (Experimental): Participants from US (aged 6 months to 17 years) received single injection of 60 μg QIV-HD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 60 µg (split-virion, inactivated)
- Group 4: Pooled QIV-SD, 15 μg (US: 6 months to 17 years) (Active Comparator): Pooled arm consisted of participants who were from US aged 6 months to 17 years, randomized to Groups 1, 2 and 3 and received single injection of 15 μg QIV-SD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: Fluarix Quadrivalent Influenza vaccine (Unadjuvanted QIV-SD) (Inactivated)
- Group 5: QIV-HD, 60 μg (Canada: 6 to <24 months) (Experimental): Participants from Canada (aged 6 to less than [<] 24 months) received single injection of 60 μg QIV-HD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 60 µg (split-virion, inactivated)
- Group 6: Adjuvanted TIV (Canada: 6 to <24 months) (Active Comparator): Participants from Canada (aged 6 to <24 months) received single injection of 7.5 μg adjuvanted TIV, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
  Interventions: Biological: FLUAD Pediatric (adjuvanted TIV) (Surface Antigen, Inactivated)

INTERVENTIONS:
Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 30 μg (split-virion, inactivated) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Arms: Group 1: QIV-HD 30 μg (US: 6 months to 17 years)
Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 45 μg, (split-virion, inactivated) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Arms: Group 2: QIV-HD 45 μg (US: 6 months to 17 years)
Biological: High-Dose Quadrivalent Influenza Vaccine (QIV-HD) 60 µg (split-virion, inactivated) — Pharmaceutical form: Suspension for injection in pre-filled syringe Route of administration: IM
  Arms: Group 3: QIV-HD, 60 μg (US: 6 months to 17 years); Group 5: QIV-HD, 60 μg (Canada: 6 to <24 months)
Biological: Fluarix Quadrivalent Influenza vaccine (Unadjuvanted QIV-SD) (Inactivated) — Pharmaceutical form: Solution for injection Route of administration: IM
  Arms: Group 4: Pooled QIV-SD, 15 μg (US: 6 months to 17 years)
Biological: FLUAD Pediatric (adjuvanted TIV) (Surface Antigen, Inactivated) — Pharmaceutical form: Solution for injection Route of administration: IM
  Arms: Group 6: Adjuvanted TIV (Canada: 6 to <24 months)

SUMMARY:
The objectives of this study were:

* To describe the safety of each dosage of high-dose quadrivalent influenza vaccine (QIV-HD) used in the study during the 28 days following each vaccination, and serious adverse events (including adverse events of special interest throughout the study).
* To describe the antibody response induced by each dosage of QIV-HD used in the study compared with unadjuvanted standard-dose quadrivalent influenza vaccine (QIV-SD) by hemagglutination inhibition (HAI) measurement method.
* To describe the antibody response induced by each dosage of QIV-HD used in the study compared with unadjuvanted QIV-SD by virus seroneutralization (SN) measurement method.
* To describe the antibody response induced by the highest acceptable dosage of QIV-HD compared with adjuvanted trivalent influenza vaccine (TIV) by HAI and virus SN measurement methods.

DETAILED DESCRIPTION:
Study duration per participant was approximately 180 days for participants who received one dose of vaccine and 208 days for participants who received two doses of vaccine.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 months to 17 years on the day of inclusion.
* Assent form was signed and dated by the participant (7 to 17 years of age) and informed consent form was signed and dated by the parent(s) or guardian(s) and by an independent witness, if required by local regulations.
* Participant and parent/guardian were able to attend all scheduled visits and complied with all study procedures.
* For participants aged <24 months: Born at full term of pregnancy (greater than or equal to [>=] 37 weeks) and/or with a birth weight >=2.5 kilogram.

Exclusion criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 3 for participants receiving 1 dose of influenza vaccine or Visit 5 for participants receiving 2 doses of influenza vaccine.
* For previously influenza vaccinated participants: Previous vaccination against influenza in the preceding 6 months with either the study vaccine or another vaccine.
* For previously influenza unvaccinated participants: Any influenza vaccination (from birth to the day of inclusion) with either the study vaccine or another influenza vaccine.
* For previously influenza unvaccinated participants: Any previous laboratory confirmed influenza infection (from birth to the day of inclusion)
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on Investigator's judgement.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >=38.0°Celsius [>=100.4°Fahrenheit]). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an immediate family member (i.e., spouse, natural or adopted child, grandchild, nephew, or niece) of the Investigator or employee with direct involvement in the proposed study.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine
* Personal history of clinically significant development delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for hepatitis B or hepatitis C.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 665 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (16):
- United States (13):
  - Investigational Site Number 8400004, San Diego, California
  - Investigational Site Number 8400001, Miami, Florida
  - Investigational Site Number 8400002, Atlanta, Georgia
  - Investigational Site Number 8400013, El Dorado, Kansas
  - Investigational Site Number 8400015, Newton, Kansas
  - Investigational Site Number 8400009, Wichita, Kansas
  - Investigational Site Number 8400007, Metairie, Louisiana
  - Investigational Site Number 8400010, Las Vegas, Nevada
  - Investigational Site Number 8400011, Warwick, Rhode Island
  - Investigational Site Number 8400003, Salt Lake City, Utah
  - Investigational Site Number 8400012, Salt Lake City, Utah
  - Investigational Site Number 8400005, Salt Lake City, Utah
  - Investigational Site Number 8400014, West Jordan, Utah
- Canada (3):
  - Investigational Site Number 1241003, Montreal
  - Investigational Site Number 1241002, Pierrefonds
  - Investigational Site Number 1241001, Québec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Chang LJ, Anderson EJ, Jeanfreau R, He Y, Hicks B, Shrestha A, Pandey A, Landolfi V, DeBruijn I; QHD04 Study Group. Safety and immunogenicity of high doses of quadrivalent influenza vaccine in children 6 months through <18 years of age: A randomized controlled phase II dose-finding trial. Vaccine. 2021 Mar 12;39(11):1572-1582. doi: 10.1016/j.vaccine.2021.02.014. Epub 2021 Feb 18. PMID 33610374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 centers in United States (US) and Canada from 09 October 2018 to 16 October 2019.
Pre-assignment Details: A total of 665 participants were enrolled in the study.
Groups:
- Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years): Participants from US (aged 6 months to 17 years) received single injection of 30 microgram (μg) high-dose quadrivalent influenza vaccine (QIV-HD), intramuscularly (IM) at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years): Pooled arm consisted of participants who were from US aged 6 months to 17 years, randomized to Groups 1, 2 and 3 and received single injection of 15 μg unadjuvanted standard-dose quadrivalent influenza vaccine (QIV-SD), IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Group 6: Adjuvanted TIV (Canada: 6 to <24 Months): Participants from Canada (aged 6 to <24 months) received single injection of 7.5 μg adjuvanted trivalent influenza vaccine (TIV), IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
Period: Overall Study
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Started | 124 | 122 | 159 | 234 | 13 | 13
Safety Analysis Set Population (SafAS) (SafAS: Included participants who had received at least one dose of the study vaccines.) | 122 | 121 | 158 | 234 | 13 | 13
Completed | 119 | 120 | 152 | 228 | 13 | 13
Not Completed | 5 | 2 | 7 | 6 | 0 | 0
Not completed — Withdrawal by parent/guardian | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 4 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the randomized participants.
Groups:
- Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years): Participants from US (aged 6 months to 17 years) received single injection of 30 μg QIV-HD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years): Pooled arm consisted of participants who were from US aged 6 months to 17 years, randomized to Groups 1, 2 and 3 and received single injection of 15 μg unadjuvanted QIV-SD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months): Participants from Canada (aged 6 to <24 months) received single injection of 60 μg QIV-HD, IM at Day 0. Participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered at Day 28.
- Total: Total of all reporting groups
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months) | Total
Number analyzed (Participants) | 124 | 122 | 159 | 234 | 13 | 13 | 665
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (3.91) | 6.1 (4.30) | 5.2 (4.22) | 5.1 (4.02) | 0.8 (0.19) | 1.0 (0.28) | 5.3 (4.13)
Age, Customized [Count of Participants; unit: Participants]
  6 - < 24 months | 0 | 0 | 0 | 0 | 13 | 13 | 26
  6 - < 36 months | 29 | 30 | 54 | 75 | 0 | 0 | 188
  36 months - < 5 years | 34 | 30 | 44 | 68 | 0 | 0 | 176
  5 - 8 years | 32 | 32 | 31 | 49 | 0 | 0 | 144
  9 - 17 years | 29 | 30 | 30 | 42 | 0 | 0 | 131
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 61 | 82 | 114 | 4 | 6 | 318
  Male | 73 | 61 | 77 | 120 | 9 | 7 | 347
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2 | 0 | 0 | 4
  Asian | 1 | 2 | 0 | 3 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 2 | 5 | 0 | 1 | 11
  Black or African American | 22 | 28 | 40 | 58 | 2 | 0 | 150
  White | 92 | 81 | 108 | 157 | 9 | 11 | 458
  More than one race | 4 | 3 | 8 | 7 | 2 | 1 | 25
  Unknown or Not Reported | 3 | 5 | 1 | 2 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AEs) After Any Vaccination
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Unsolicited AEs includes both serious (SAEs) and non-serious unsolicited AEs. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. All participants were observed for 30 minutes after vaccination, and any unsolicited systemic AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes after any vaccination
Population: Analysis was performed on SafAS population which included participants who had received at least one dose of the study vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 122 | 121 | 158 | 234 | 13 | 13
Participants | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited Adverse Events After Any Vaccination
Description: An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset window post-vaccination. Unsolicited AEs included both serious and non-serious unsolicited AEs. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. Adverse reactions (ARs) were AEs related to vaccination. An injection site reaction was an AR at and around the injection site. Systemic AEs were all AEs that were not injection or administration site reactions.
Time Frame: Within 28 days after any vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 122 | 121 | 158 | 234 | 13 | 13
Participants
  Unsolicited AE | 46 | 46 | 53 | 80 | 11 | 12
  Unsolicited non-serious AR | 4 | 8 | 8 | 10 | 1 | 3
  Unsolicited non-serious injection site AR | 0 | 3 | 0 | 0 | 0 | 1
  Unsolicited non-serious systemic AE | 46 | 45 | 52 | 80 | 11 | 12
  Unsolicited non-serious systemic AR | 4 | 5 | 8 | 10 | 1 | 2

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) After Any Vaccination
Description: An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An SAE which caused death of the participant was considered as fatal SAE. Adverse events of special interest (AESIs) were defined as SAEs which included new onset of Guillain-Barré syndrome, encephalitis/myelitis (including transverse myelitis), Bell's palsy, convulsions, optic neuritis, and brachial neuritis.
Time Frame: From Day 0 up to 6 months (i.e. 180 days) post last vaccination
Population: Analysis was performed on the SafAS population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 122 | 121 | 158 | 234 | 13 | 13
Participants
  SAE | 0 | 0 | 2 | 0 | 0 | 1
  Fatal SAE | 0 | 0 | 0 | 0 | 0 | 0
  AESI | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Achieving Seroconversion Against Antigens Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: Anti-influenza antibodies were measured by hemagglutination inhibition (HAI) assay for strains A/H1N1, A/H3N2, B/Victoria and B/Yamagata lineage. Seroconversion: defined as either HAI titer <10(1/dilution) at Day 0 and post-vaccination titer greater than or equal to (>=)40(1/dilution) at Day 28, or HAI titer >=10(1/dilution) at Day 0 and >=4-fold increase in HAI titer (1/dilution) at Day 28. Data for this Outcome Measure (OM) was planned to be collected and reported for dose level (QIV-HD 30μg and 45μg) matched separate groups for QIV-SD (Groups 4a, 4b and 4c), instead of pooled QIV-SD arm. Due to complex study design and analysis of doses and age groups, QIV-SD group participants, who matched to participants in QIV-HD 30μg and 45μg dose formulations groups (who were 9 through 17 years old and shared matching age group with QIV-SD control group), included in Groups 4a, 4b and 4c in this OM might be counted in more than once in QIV-SD arms for different dose levels, as applicable.
Time Frame: Day 28 post any vaccination
Population: Analysis was performed on immunogenicity analysis set (IAS) population which included randomized participants who received 1 dose or 2 doses of study vaccine and had a post-vaccination blood sample. Here, 'number analyzed' = number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Groups:
- Group 4a: QIV-SD, 15 μg, (US: 6 Months to 17 Years): Participants from US (aged 6 months to 17 years) received 15 μg QIV-SD, IM and were restricted for comparison to relevant experimental study group QIV-HD 30 μg.
- Group 4b: QIV-SD, 15 μg, (US: 6 Months to 17 Years): Participants from US (aged 6 months to 17 years) received 15 μg QIV-SD, IM and were restricted for comparison to relevant experimental study group QIV-HD 45 μg.
- Group 4c: QIV-SD, 15 μg, (US: 6 Months to 17 Years): Participants from US (aged 6 months to 17 years) received 15 μg QIV-SD, IM and were restricted for comparison to relevant experimental study group QIV-HD 60 μg.
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4a: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 4b: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 4c: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 40 | 41 | 157 | 13 | 13
Participants
  A/H1N1: number analyzed (Participants) | 110 | 112 | 141 | 39 | 41 | 148 | 11 | 12
  A/H1N1 | 72 | 71 | 107 | 26 | 24 | 98 | 8 | 11
  A/H3N2: number analyzed (Participants) | 109 | 111 | 140 | 38 | 41 | 146 | 11 | 12
  A/H3N2 | 63 | 79 | 102 | 18 | 20 | 71 | 8 | 12
  B/Victoria: number analyzed (Participants) | 110 | 111 | 141 | 39 | 41 | 148 | 11 | 12
  B/Victoria | 84 | 94 | 117 | 28 | 30 | 111 | 6 | 12
  B/Yamagata: number analyzed (Participants) | 110 | 109 | 141 | 38 | 41 | 147 | 11 | 12
  B/Yamagata | 79 | 85 | 120 | 26 | 31 | 117 | 8 | 1

5. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Antibodies Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: GMTs of anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage. Data for this OM was planned to be collected and reported for dose level (QIV-HD 30 μg and QIV-HD 45 μg) matched separate groups for QIV-SD (Groups 4a, 4b and 4c), instead of pooled QIV-SD arm. Due to the complex study design and analysis of the dose formulation and age groups in the study, QIV-SD group participants, who matched to participants in the QIV-HD 30 μg and QIV-HD 45 μg dose formulations groups (who were 9 through 17 years old and shared a matching age group with QIV-SD control group), included in Groups 4a, 4b and 4c in this OM might be counted in more than once in QIV-SD arms for different dose levels, as applicable.
Time Frame: Day 28 post any vaccination
Population: Analysis was performed on IAS population. Here, 'number analyzed' = number of participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4a: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 4b: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 4c: QIV-SD, 15 μg, (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 40 | 41 | 157 | 13 | 13
titers (1/dilution)
  A/H1N1: number analyzed (Participants) | 116 | 114 | 145 | 40 | 41 | 151 | 13 | 12
  A/H1N1 | 673 [525 to 863] | 676 [524 to 873] | 834 [674 to 1033] | 698 [419 to 1161] | 791 [480 to 1303] | 618 [461 to 830] | 59.7 [27.0 to 132] | 604 [261 to 1398]
  A/H3N2: number analyzed (Participants) | 116 | 113 | 144 | 39 | 41 | 151 | 13 | 12
  A/H3N2 | 518 [399 to 671] | 781 [600 to 1017] | 770 [604 to 982] | 314 [184 to 538] | 441 [264 to 738] | 307 [239 to 395] | 66.4 [33.0 to 133] | 604 [386 to 946]
  B/Victoria: number analyzed (Participants) | 116 | 113 | 145 | 40 | 41 | 151 | 13 | 12
  B/Victoria | 378 [296 to 483] | 432 [334 to 560] | 494 [400 to 612] | 296 [194 to 452] | 468 [302 to 726] | 310 [246 to 390] | 56.6 [26.2 to 122] | 1244 [767 to 2016]
  B/Yamagata: number analyzed (Participants) | 116 | 112 | 144 | 39 | 41 | 151 | 13 | 12
  B/Yamagata | 723 [582 to 899] | 720 [556 to 932] | 877 [722 to 1066] | 706 [474 to 1050] | 727 [501 to 1054] | 580 [466 to 721] | 75.8 [38.9 to 148] | 21.8 [12.3 to 38.6]

6. Primary Outcome: Geometric Mean Titer Ratios (GMTRs) of Influenza Antibodies Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: GMTs of anti-influenza antibodies were measured using an HAI assay for 4 strains: A/H1N1, A/H3N2, B Victoria lineage, and B Yamagata lineage. GMTRs were calculated as the ratio of GMTs post-vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28 (post any vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
ratio
  A/H1N1: Day 28/Day 0: number analyzed (Participants) | 110 | 112 | 141 | 217 | 11 | 12
  A/H1N1: Day 28/Day 0 | 8.55 [6.39 to 11.4] | 10.0 [7.31 to 13.7] | 16.3 [12.1 to 22.0] | 10.1 [8.07 to 12.8] | 1.41 [0.878 to 2.28] | 4.76 [2.72 to 8.32]
  A/H3N2: Day 28/Day 0: number analyzed (Participants) | 109 | 111 | 140 | 214 | 11 | 12
  A/H3N2: Day 28/Day 0 | 6.42 [4.95 to 8.34] | 9.35 [7.15 to 12.2] | 10.3 [8.09 to 13.0] | 4.61 [3.90 to 5.45] | 1.41 [1.00 to 2.00] | 15.5 [8.89 to 27.2]
  B/Victoria: Day 28/Day 0: number analyzed (Participants) | 110 | 111 | 141 | 217 | 11 | 12
  B/Victoria: Day 28/Day 0 | 10.7 [8.31 to 13.7] | 11.7 [9.30 to 14.7] | 16.7 [13.2 to 21.0] | 11.0 [9.24 to 13.2] | 1.37 [0.949 to 1.98] | 11.0 [6.28 to 19.2]
  B/Yamagata: Day 28/Day 0: number analyzed (Participants) | 110 | 109 | 141 | 215 | 11 | 12
  B/Yamagata: Day 28/Day 0 | 9.28 [7.10 to 12.1] | 11.4 [8.83 to 14.7] | 18.1 [13.9 to 23.6] | 9.77 [8.15 to 11.7] | 1.71 [1.07 to 2.73] | 0.944 [0.785 to 1.13]

7. Primary Outcome: Number of Participants With Neutralization Antibody Titers >= 40 (1/Dilution) Following Vaccination With Either a High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: GMT was measured for each influenza strain using HAI assay method for 4 strains: A/H1N1, A/H3N2, B/Victoria lineage, and B/Yamagata lineage.
Time Frame: Day 28 post any vaccination
Population: Analysis was performed on the IAS population. Here, 'number analyzed' = number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
Participants
  A/H1N1: Day 28: number analyzed (Participants) | 116 | 114 | 145 | 221 | 13 | 12
  A/H1N1: Day 28 | 113 | 110 | 142 | 198 | 0 | 7
  A/H3N2: Day 28: number analyzed (Participants) | 116 | 113 | 144 | 220 | 13 | 12
  A/H3N2: Day 28 | 111 | 110 | 139 | 198 | 0 | 9
  B/Victoria: Day 28: number analyzed (Participants) | 116 | 113 | 145 | 221 | 13 | 12
  B/Victoria: Day 28 | 112 | 108 | 140 | 202 | 0 | 9
  B/Yamagata: Day 28: number analyzed (Participants) | 116 | 112 | 144 | 220 | 13 | 12
  B/Yamagata: Day 28 | 115 | 109 | 142 | 215 | 1 | 1

8. Primary Outcome: Geometric Mean Titers of Influenza Antibodies (Measured by Seroneutralization [SN] Assay) Following Vaccination With Either High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: GMT was measured for each influenza strain using SN assay method for 4 strains: A/H1N1, A/H3N2, B/Victoria lineage, and B/Yamagata lineage.
Time Frame: Day 28 post any vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
titers (1/dilution)
  A/H1N1: number analyzed (Participants) | 112 | 112 | 147 | 216 | 12 | 11
  A/H1N1 | 6589 [4959 to 8754] | 6213 [4672 to 8264] | 7045 [5514 to 9001] | 4948 [3676 to 6659] | 33.8 [14.8 to 76.9] | 234 [32.0 to 1708]
  A/H3N2: number analyzed (Participants) | 113 | 111 | 142 | 215 | 11 | 11
  A/H3N2 | 641 [515 to 798] | 921 [718 to 1181] | 884 [717 to 1091] | 411 [347 to 487] | 54.4 [35.3 to 83.9] | 188 [119 to 298]
  B/Victoria: number analyzed (Participants) | 113 | 112 | 146 | 216 | 12 | 11
  B/Victoria | 500 [375 to 667] | 605 [444 to 825] | 628 [484 to 815] | 378 [302 to 472] | 6.05 [4.54 to 8.07] | 57.9 [39.5 to 84.9]
  B/Yamagata: number analyzed (Participants) | 112 | 112 | 146 | 214 | 12 | 11
  B/Yamagata | 1147 [893 to 1474] | 1159 [865 to 1552] | 1254 [1015 to 1549] | 846 [698 to 1026] | 17.6 [11.1 to 27.8] | 17.4 [9.86 to 30.6]

9. Primary Outcome: Geometric Mean Titers Ratio of Influenza Antibodies (Measured by Seroneutralization Assay) Following Vaccination With Either High-Dose Quadrivalent Influenza Vaccine or Standard-Dose Quadrivalent Influenza Vaccine or Adjuvanted Trivalent Influenza Vaccine
Description: GMTRs of anti-influenza antibodies were measured using SN assay method for 4 strains: A/H1N1, A/H3N2, B/Victoria lineage and B/Yamagata lineage. GMTRs were calculated as the ratio of GMTs post vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination), Day 28 (post any vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
ratio
  A/H1N1: Day 28/Day 0: number analyzed (Participants) | 103 | 105 | 138 | 206 | 10 | 11
  A/H1N1: Day 28/Day 0 | 11.3 [7.67 to 16.7] | 18.8 [12.1 to 29.4] | 29.1 [19.6 to 43.2] | 14.5 [11.0 to 19.0] | 2.38 [0.663 to 8.53] | 7.12 [3.00 to 16.9]
  A/H3N2: Day 28/Day 0: number analyzed (Participants) | 101 | 101 | 134 | 206 | 10 | 11
  A/H3N2: Day 28/Day 0 | 3.60 [2.98 to 4.34] | 5.20 [4.11 to 6.59] | 5.54 [4.58 to 6.70] | 2.66 [2.34 to 3.04] | 1.04 [0.629 to 1.72] | 2.81 [1.65 to 4.78]
  B/Victoria: Day 28/Day 0: number analyzed (Participants) | 102 | 105 | 137 | 205 | 10 | 11
  B/Victoria: Day 28/Day 0 | 12.4 [9.51 to 16.2] | 15.4 [11.9 to 20.0] | 19.9 [15.1 to 26.3] | 12.7 [10.4 to 15.4] | 1.03 [0.612 to 1.74] | 10.5 [6.73 to 16.3]
  B/Yamagata: Day 28/Day 0: number analyzed (Participants) | 101 | 103 | 137 | 204 | 10 | 11
  B/Yamagata: Day 28/Day 0 | 9.75 [7.50 to 12.7] | 11.5 [9.06 to 14.7] | 14.1 [11.1 to 17.8] | 8.49 [7.18 to 10.0] | 1.16 [0.604 to 2.24] | 1.10 [0.760 to 1.61]

10. Primary Outcome: Number of Participants With Neutralization Antibody Titers Above Pre-Defined Thresholds
Description: Neutralizing Antibody titer was measured for each influenza strain with SN assay method for 4 strains: A/H1N1, A/H3N2, B/Victoria lineage, and B/Yamagata lineage at pre-defined thresholds of >=20, >=40 and >=80 (1/dilution).
Time Frame: Day 28 post any vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
Participants
  A/H1N1: >=20 (1/dilution): number analyzed (Participants) | 112 | 112 | 147 | 216 | 13 | 11
  A/H1N1: >=20 (1/dilution) | 112 | 112 | 147 | 208 | 13 | 11
  A/H1N1: >=40 (1/dilution): number analyzed (Participants) | 112 | 112 | 147 | 216 | 13 | 11
  A/H1N1: >=40 (1/dilution) | 112 | 112 | 147 | 202 | 12 | 11
  A/H1N1: >=80 (1/dilution): number analyzed (Participants) | 112 | 112 | 147 | 216 | 13 | 11
  A/H1N1: >=80 (1/dilution) | 111 | 111 | 146 | 201 | 11 | 11
  A/H3N2: >=20 (1/dilution): number analyzed (Participants) | 113 | 111 | 142 | 215 | 13 | 11
  A/H3N2: >=20 (1/dilution) | 113 | 111 | 142 | 214 | 13 | 11
  A/H3N2: >=40 (1/dilution): number analyzed (Participants) | 113 | 111 | 142 | 215 | 13 | 11
  A/H3N2: >=40 (1/dilution) | 111 | 111 | 141 | 208 | 13 | 11
  A/H3N2: >=80 (1/dilution): number analyzed (Participants) | 113 | 111 | 142 | 215 | 13 | 11
  A/H3N2: >=80 (1/dilution) | 107 | 107 | 138 | 190 | 11 | 11
  B/Victoria: >=20 (1/dilution): number analyzed (Participants) | 113 | 112 | 146 | 216 | 13 | 11
  B/Victoria: >=20 (1/dilution) | 110 | 108 | 143 | 201 | 9 | 11
  B/Victoria: >=40 (1/dilution): number analyzed (Participants) | 113 | 112 | 146 | 216 | 13 | 11
  B/Victoria: >=40 (1/dilution) | 108 | 104 | 136 | 195 | 8 | 11
  B/Victoria: >=80 (1/dilution): number analyzed (Participants) | 113 | 112 | 146 | 216 | 13 | 11
  B/Victoria: >=80 (1/dilution) | 99 | 99 | 128 | 181 | 6 | 11
  B/Yamagata: >=20 (1/dilution): number analyzed (Participants) | 112 | 112 | 146 | 214 | 13 | 11
  B/Yamagata: >=20 (1/dilution) | 111 | 112 | 146 | 213 | 13 | 10
  B/Yamagata: >=40 (1/dilution): number analyzed (Participants) | 112 | 112 | 146 | 214 | 13 | 11
  B/Yamagata: >=40 (1/dilution) | 111 | 108 | 145 | 208 | 9 | 6
  B/Yamagata: >=80 (1/dilution): number analyzed (Participants) | 112 | 112 | 146 | 214 | 13 | 11
  B/Yamagata: >=80 (1/dilution) | 110 | 103 | 140 | 201 | 7 | 2

11. Primary Outcome: Number of Participants With Two-Fold and Four-Fold Increase in Neutralization Antibody Titer
Description: Neutralizing Antibody titer was measured for each influenza strain with SN method for 4 strains: A/H1N1, A/H3N2, B/Victoria lineage, and B/Yamagata lineage. 2-fold and 4-fold rise was defined as the computed value = post-vaccination computed value / pre-vaccination computed value.
Time Frame: Day 28 post any vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 118 | 115 | 156 | 227 | 13 | 13
Participants
  2-Fold Rise: A/H1N1: number analyzed (Participants) | 103 | 105 | 138 | 206 | 10 | 11
  2-Fold Rise: A/H1N1 | 80 | 83 | 118 | 168 | 6 | 10
  4-Fold Rise: A/H1N1: number analyzed (Participants) | 103 | 105 | 138 | 206 | 10 | 11
  4-Fold Rise: A/H1N1 | 65 | 70 | 104 | 141 | 5 | 9
  2-Fold Rise: A/H3N2: number analyzed (Participants) | 101 | 101 | 134 | 206 | 10 | 11
  2-Fold Rise: A/H3N2 | 69 | 77 | 110 | 111 | 2 | 7
  4-Fold Rise: A/H3N2: number analyzed (Participants) | 101 | 101 | 134 | 206 | 10 | 11
  4-Fold Rise: A/H3N2 | 44 | 51 | 72 | 61 | 0 | 3
  2-Fold Rise: B/Victoria: number analyzed (Participants) | 102 | 105 | 137 | 205 | 10 | 11
  2-Fold Rise: B/Victoria | 95 | 99 | 131 | 185 | 2 | 11
  4-Fold Rise: B/Victoria: number analyzed (Participants) | 102 | 105 | 137 | 205 | 10 | 11
  4-Fold Rise: B/Victoria | 80 | 88 | 113 | 158 | 0 | 10
  2-Fold Rise: B/Yamagata: number analyzed (Participants) | 101 | 103 | 137 | 204 | 10 | 11
  2-Fold Rise: B/Yamagata | 84 | 95 | 127 | 187 | 4 | 3
  4-Fold Rise: B/Yamagata: number analyzed (Participants) | 101 | 103 | 137 | 204 | 10 | 11
  4-Fold Rise: B/Yamagata | 71 | 81 | 109 | 142 | 1 | 0

12. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the administered vaccination. Solicited injection site reactions included tenderness/pain, erythema, swelling, induration and bruising.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed on the SafAS population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 122 | 119 | 158 | 232 | 13 | 13
Participants
  Injection site tenderness/pain | 81 | 84 | 100 | 116 | 6 | 5
  Injection site erythema | 31 | 30 | 40 | 48 | 5 | 8
  Injection site swelling | 17 | 15 | 34 | 23 | 2 | 2
  Injection site induration | 21 | 18 | 26 | 22 | 4 | 5
  Injection site bruising | 10 | 10 | 13 | 16 | 1 | 2

13. Primary Outcome: Number of Participants With Solicited Systemic Reactions After Any Vaccination
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the administered vaccination. Solicited systemic reactions included fever, vomiting, crying abnormal, drowsiness, appetite loss and irritability. Fever was planned to be evaluated for the whole population where as, the other events (vomiting, crying abnormal, drowsiness, appetite lost, and irritability) were planned to be evaluated only in the participants aged 6 months to <36 months.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed on the SafAS population. Here, 'number analyzed' = number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
Number analyzed (Participants) | 122 | 121 | 158 | 234 | 13 | 13
Participants
  Fever: number analyzed (Participants) | 122 | 120 | 158 | 231 | 13 | 13
  Fever | 5 | 6 | 15 | 11 | 5 | 6
  Vomiting: number analyzed (Participants) | 29 | 30 | 54 | 74 | 13 | 13
  Vomiting | 1 | 2 | 7 | 11 | 5 | 7
  Crying abnormal: number analyzed (Participants) | 29 | 30 | 54 | 74 | 13 | 13
  Crying abnormal | 11 | 9 | 10 | 20 | 6 | 9
  Drowsiness: number analyzed (Participants) | 29 | 30 | 54 | 74 | 13 | 13
  Drowsiness | 14 | 11 | 12 | 17 | 5 | 5
  Appetite lost: number analyzed (Participants) | 29 | 30 | 54 | 74 | 13 | 13
  Appetite lost | 6 | 10 | 15 | 20 | 11 | 11
  Irritability: number analyzed (Participants) | 29 | 30 | 54 | 74 | 13 | 13
  Irritability | 14 | 13 | 18 | 23 | 6 | 12

14. Primary Outcome: Number of Participants With Solicited Systemic Reactions After Any Vaccination: Participants Aged >36 Months
Description: A solicited reaction was an expected adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) prelisted (i.e., solicited) in the CRB and considered as related to the administered vaccination. Solicited systemic reactions included: headache, malaise, myalgia and shivering.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed on the SafAS population. Here, "overall number of participants analyzed"= participants evaluable for this outcome measure. Data not collected and reported for Groups 5 and 6 because none of the participants in both groups lies in the age group of >36 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years)
Number analyzed (Participants) | 93 | 89 | 104 | 158
Participants
  Headache | 18 | 18 | 22 | 21
  Malaise | 16 | 28 | 27 | 32
  Myalgia | 29 | 30 | 32 | 42
  Shivering | 1 | 8 | 8 | 6

ADVERSE EVENTS:
Time Frame: AEs were collected from Day 0 (post-vaccination) up to 28 days after last vaccination. Solicited Reaction (SR) data were collected up to Day 7 after any vaccination. SAE data were collected throughout the study (up to 180 days after last vaccination).
Description: An SR was an AE that was prelisted (i.e., solicited) in the CRB and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRB in terms of diagnosis and/or onset window post-vaccination. Analysis was performed on SafAS population.
Arm/Group | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months)
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/121 | 0/158 | 0/234 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/121 | 2/158 | 0/234 | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 101/122 | 100/121 | 118/158 | 165/234 | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) (N=122) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) (N=121) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) (N=158) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) (N=234) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) (N=13) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months) (N=13)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: QIV-HD 30 μg (US: 6 Months to 17 Years) (N=122) | Group 2: QIV-HD 45 μg (US: 6 Months to 17 Years) (N=121) | Group 3: QIV-HD, 60 μg (US: 6 Months to 17 Years) (N=158) | Group 4: Pooled QIV-SD, 15 μg (US: 6 Months to 17 Years) (N=234) | Group 5: QIV-HD, 60 μg (Canada: 6 to <24 Months) (N=13) | Group 6: Adjuvanted TIV (Canada: 6 to <24 Months) (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (6) | 9 (10) | 12 (13) | 1 (1) | 4 (8)
Oral Mucosal Eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (12) | 10 (10) | 12 (13) | 15 (16) | 5 (9) | 7 (9)
Chills (General disorders) | 1 (1) | 8 (8) | 8 (8) | 6 (6) | 0 (0) | 0 (0)
Crying (General disorders) | 11 (12) | 9 (10) | 10 (12) | 20 (24) | 6 (9) | 9 (10)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Bruising (General disorders) | 10 (10) | 11 (11) | 13 (14) | 16 (16) | 1 (1) | 2 (2)
Injection Site Erythema (General disorders) | 31 (32) | 30 (32) | 40 (44) | 48 (52) | 5 (7) | 8 (9)
Injection Site Induration (General disorders) | 21 (22) | 19 (20) | 26 (27) | 22 (24) | 4 (5) | 5 (6)
Injection Site Pain (General disorders) | 81 (89) | 84 (96) | 100 (111) | 116 (126) | 6 (8) | 5 (6)
Injection Site Swelling (General disorders) | 17 (17) | 15 (17) | 34 (35) | 23 (25) | 2 (2) | 2 (2)
Injection Site Warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 16 (16) | 28 (29) | 27 (27) | 32 (33) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (12) | 10 (11) | 19 (22) | 24 (25) | 9 (15) | 9 (17)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (4) | 3 (4)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 8 (8) | 5 (5) | 7 (9) | 7 (13)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 0 (0) | 6 (6) | 8 (8) | 0 (0) | 1 (1)
Tongue Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 10 (11) | 15 (18) | 20 (24) | 11 (14) | 11 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (33) | 30 (31) | 33 (34) | 43 (45) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 18 (19) | 19 (19) | 22 (22) | 22 (22) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 14 (15) | 11 (12) | 12 (17) | 18 (21) | 5 (6) | 5 (7)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 14 (16) | 13 (15) | 18 (24) | 23 (27) | 7 (11) | 12 (19)
Sleep Terror (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 19 (22) | 15 (17) | 30 (30) | 2 (4) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 4 (7) | 13 (13) | 0 (0) | 1 (1)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT03698279/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03698279/SAP_001.pdf